CLINICAL TRIAL: NCT03593460
Title: Phase II, Open Label, Adaptive Design, Multiple Dose Finding Study to Investigate Synthetic PreImplantation Factor (sPIF) in Patients With Autoimmune Hepatitis (AIH)
Brief Title: Phase II AutoImmune Hepatitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: BioIncept changed the focus of future drug development
Sponsor: Christopher O'Brien, MD (Other)
Collaborators: BioIncept LLC (Industry)
Responsible Party: Sponsor-Investigator, Christopher O'Brien, MD, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: sPIF-US-AIH-002
Record Dates: First submitted 2018-06-07; First posted 2018-07-20 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis, Autoimmune
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — preimplantation factor, synthetic

STUDY DESIGN:
Intervention Model Description: Adaptive Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- sPIF 1 mg/kg (Starting Dose) (Experimental): Patients will be administered a starting dose of sPIF 1mg/kg (n=10/cohort) for 14 days assessing safety, tolerability and clinical response based on the effect on ALT levels
  Interventions: Drug: Synthetic PreImplantation Factor
- sPIF 2 mg/kg (Experimental): Patients will be dosed at 2mg/kg sPIF for 14 days assessing safety, tolerability and clinical response based on the effect on ALT levels.
  Interventions: Drug: Synthetic PreImplantation Factor
- sPIF 3 mg/kg (Experimental): Patients will be administered a starting dose of sPIF 3mg/kg (n=10/cohort) for 14 days assessing safety, tolerability and clinical response based on the effect on ALT levels
  Interventions: Drug: Synthetic PreImplantation Factor
- sPIF 4 mg/kg (Experimental): Patients will be administered a starting dose of sPIF 4mg/kg (n=10/cohort) for 14 days assessing safety, tolerability and clinical response based on the effect on ALT levels
  Interventions: Drug: Synthetic PreImplantation Factor
- sPIF 5 mg/kg (Experimental): Patients will be administered a starting dose of sPIF 5mg/kg (n=10/cohort) for 14 days assessing safety, tolerability and clinical response based on the effect on ALT levels.
  Interventions: Drug: Synthetic PreImplantation Factor

INTERVENTIONS:
Drug: Synthetic PreImplantation Factor — peptide
  Other Names: sPIF

SUMMARY:
This is a Phase IIa open label adaptive design dose finding study in male and female patients with autoimmune hepatitis (AIH) with compensated liver function currently under standard of care. The purpose of this study is to evaluate the sPIF dose that normalizes and maintains the serum ALT when given for 14 doses.

Autoimmune Hepatitis is disease where the patient's immune system produces an inappropriate immune response against their own liver. PreImplantation factor (PIF) is a substance that is secreted by viable fetuses during pregnancy. PIF initiates both maternal tolerance preventing the loss/rejection of the fetus. Synthetic PIF (sPIF) successfully translates PIF endogenous properties to pregnant and non-pregnant immune disorders. sPIF was found to be effective in preclinical models of autoimmunity and transplantation. Specifically, sPIF protected the liver against immune attack.

DETAILED DESCRIPTION:
The study is an open label, dose finding trial in patients with AIH who have an elevated ALT levels. Patients will be administered a starting dose of sPIF 1mg/kg (n=10/cohort) for 14 days assessing safety, tolerability and clinical response based on the effect on ALT levels until day 84. This will be followed by enrolling (n=10) patients administering 2mg/kg sPIF for 14 days assessing safety, tolerability and clinical response based on the effect on ALT levels until day 84. This be followed by an interim analysis that will determine clinical efficacy by comparing the 1mg and 2mg dose results; testing the decrease in mean ALT percent and determining the number of patients in remission defined as normalized ALT level. The successful cohort will enroll additional patients to enable power analysis. If no significant improvement is observed in the two cohorts, N=10 patients will be enrolled and administered 3mg/kg sPIF for 14 days assessing safety and tolerability. If no significant improvement is noted and safety and tolerability is maintained additional 10 patients will be enrolled at 4mg/kg. Following the same analysis, the maximal dose to be administered will be 5mg/kg.

ELIGIBILITY:
Written informed consent must be obtained before any assessment is performed. Patients with a confirmed diagnosis of AIH either Type II or Type II, based on the International Criteria for the Diagnosis of AIH, will be enrolled at screening.

* Males and females aged from 18 to 75 years old, of non-child bearing potential
* Females must be either:

Postmenopausal for greater than two years Postmenopausal for less than two years with an FSH level greater > 40mIU/mL Documented as surgically sterile (bilateral tubal ligation, bilateral oophorectomy or post-hysterectomy) at least three months prior to the screening evaluation Or be greater than age 40, does not want more children, is currently using at least one effective method of birth control at the time of screening and agrees to using two effective methods of birth control starting with Study day 0 and through the 42 days duration of the study

• Must have in the judgment of the Investigator, the diagnosis of AIH, or have a score on the International Criteria for the Diagnosis of AIH (Appendix 2) of: Pretreatment score ≥15 Post-treatment score of ≥17

* Treatment with prednisone and/or other oral, immunosuppressive drug(s) must be stabilized for 6 weeks prior to screening for this study.
* All patients with an abnormal ALT confirmed by two measurements 2 weeks apart at screening, with the present dose(s) of their immunosuppressant medication(s)
* Patients do not have to have a documented relapse after completion of an initial course of therapy
* Permitted concomitant immunosuppressant medications will include:

Azathioprine dose equal to/or less 100 mg per day Budesonide dose equal to/or less 9 mg per day Mycophenolate metil equal to/or less 3000 mg per day Prednisone equal to/or less than 30 mg per day Ursodeoxycholic acid equal to/or less than 1500 mg er day Prograf equal to/or less than 6 mg per day

* Patients must agree to abstain from alcohol and illicit drugs use during their participation in the study protocol
* ALT and AST levels greater than 2 times less than five times the upper limit of the normal (reference) range (ULN) and have no clinical or laboratory evidence of hepatic decompensation (i.e., platelets ≥ 100,000/mm, total bilirubin ≤ 1.5 × ULN, prothrombin time ≤ 1.2 × ULN and albumin ≥ 3.0 g/dL) for inclusion.
* Normal renal function as determined by a serum creatinine

Exclusion criteria

Patients fulfilling any of the following criteria are not eligible for inclusion in this study. No additional exclusions may be applied by the Investigator, to ensure that the study population will be representative of all eligible patients.

* Any other forms of chronic liver disease that is not under treatment
* Decompensated liver disease defined on the basis of any one of the following laboratory parameters at the screening evaluation: total bilirubin > 1.5 × ULN, prothrombin time > 1.2 × ULN, platelets ≤ 100,000/mm3, or albumin < 3 g/dL OR current or prior history of clinical hepatic decompensation (e.g., ascites, jaundice, encephalopathy or variceal hemorrhage)
* Hemoglobin < 11 g/dL at the screening evaluation
* Serological evidence of infection with HIV upon review of the medical record
* Evidence of hepatocellular carcinoma (i.e., screening α-fetoprotein > 50 ng/mL or other standard of care measure and ultrasound)
* Patients with, or a history of clinically significant oncologic, pulmonary, hepatic, gastrointestinal, renal, other cardiovascular, hematologic, metabolic, endocrine, neurologic, immunologic or hematologic illness or any other major medical disorder that, in the judgment of the Investigator, would interfere with patient treatment, assessment or compliance with the protocol or should otherwise preclude their participation in this trial
* Have received therapy with potentially hepatotoxic drugs within 3 months (90 days) prior to day 1 or are expected to receive such therapy during the study
* Patients who are expected to receive a change in their immunosuppressant therapies during the protocol
* Patients who may receive chemotherapeutic agents (e.g. immunoglobulins and other immune- or cytokine-based therapies) during the study for any other medical condition
* Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days until the expected pharmacodynamic effect has returned to baseline, whichever is longer
* History of hypersensitivity to study drug or its excipients
* Hepatitis B and C, infectious hepatitis (documented in medical record may need to repeat prior to enrollment)
* Tuberculosis (documented in medical record)
* Primary sclerosing cholangitis, primary biliary cholangitis (documented in medical record and may need to repeat prior to enrollment)
* Alpha-1 antitrypsin deficiency, hemochromatosis, or Wilson's disease (documented in the medical record)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of multiple ascending, subcutaneously administered doses of sPIF in patients with autoimmune hepatitis (AIH) by measuring changes in ALT | 12 weeks
  Change of ALT from baseline to normal range
Evaluate the pharmacokinetics of sPIF levels in the circulation after multiple ascending, subcutaneously administered doses of sPIF by normalization of liver enzymes, immunoglobulins, and bilirubin levels | 12 weeks
  normalized AST, ALP, GGT, IgG, and bilirubin levels
Evaluate the safety and tolerability of the increased sPIF dose and treatment duration by no SAEes greater than grade 3 | 12 weeks
  No SAE > Grade 3 observed

OTHER OUTCOMES:
Determine the proportion of patients achieving total remission by normalization of serum ALT levels | 12 weeks
  Normalization in serum ALT levels (Males <45U/L and females <30 U/L)
Determine the proportion of patients achieving partial remission by obervation of ALT levels greater than 1 but less than 2 the upper limit of normal | 12 weeks
  ALT levels > 1x ULN and <2x ULN

CONTACTS AND LOCATIONS:
Overall Officials: eytan barnea, MD, Principal Investigator — BioIncept LLC

REFERENCES:
- [Result] Barnea ER, Rambaldi M, Paidas MJ, Mecacci F. Reproduction and autoimmune disease: important translational implications from embryo-maternal interaction. Immunotherapy. 2013 Jul;5(7):769-80. doi: 10.2217/imt.13.59. PMID 23829627